CLINICAL TRIAL: NCT03799198
Title: Real World Effectiveness of Combining an Employer-based Weight Management Program With Medication for Chronic Weight Management in Employees With Obesity - a Pragmatic Randomized Trial
Brief Title: Real World Effectiveness of Combining an Employer-based Weight Management Program With Medication for Chronic Weight Management in Employees With Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8022-4432; U1111-1218-8104 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WMP + Rx (Experimental): Participants will receive Cleveland Clinic's Integrated Medical WMP with medication for chronic weight management (Rx) for approximately one year. After discussing with the study doctor, participants will receive one of the following listed 5 drugs approved by the Food and Drug Administration (FDA) for long-term weight loss: 1) orlistat, 2) lorcaserin or lorcaserin extended-release, 3) phentermine/topiramate extended-release, 4) naltrexone/bupropion extended-release and 5) liraglutide 3.0 mg.
  Interventions: Other: Weight Management Program (WMP); Drug: Medication for chronic weight management (Rx)
- WMP alone (Active Comparator): Participants will receive Cleveland Clinic's Integrated Medical WMP alone for approximately one year.
  Interventions: Other: Weight Management Program (WMP)

INTERVENTIONS:
Other: Weight Management Program (WMP) — As part of usual care, participants will: 1) Discuss and choose one of three diet options: protein-sparing modified fast, Mediterranean, or meal replacement. 2) Be referred to a nutritionist appointment. 3) Initiate a series of twelve monthly study visits in the context of shared medical appointments (SMAs) covering nutrition, physical activity, appetite control, sleep issues, and anxiety/depression/stress. 4) Be referred to an exercise physiologist for a personalized physical activity program. 5) If assessed relevant by the study clinician, be referred to a mental health specialist and/or sleep clinic.
Drug: Medication for chronic weight management (Rx) — Following listed 5 drugs will be administered as prescribed by the study doctor:
  1) Orlistat (Xenical® pills, per os [p.o.; by mouth]). 2) Lorcaserin or lorcaserin extended-release (Belviq®/Belviq XR® pills, p.o.). 3) Phentermine/topiramate extended-release (Qsymia® pills, p.o.). 4) Naltrexone/bupropion extended-release (Contrave® pills, p.o.). 5) Liraglutide 3.0 mg (Saxenda® injections, subcutaneously [under the skin]).
  Arms: WMP + Rx

SUMMARY:
Researchers are doing this study to compare the effects of drugs approved for long-term weight loss combined with an employer-based weight management program with the effects of the weight management program without drugs for weight loss. If participants agree to be in this study, they will join the Cleveland Clinic Integrated Medical Weight Management Program (WMP). Participants will be assigned by chance (like flipping a coin) to one of two treatment groups: A) Group 1: Cleveland Clinic Integrated Medical WMP + medication for long-term weight loss. B) Group 2: Cleveland Clinic Integrated Medical WMP without medication for weight loss. Participants have an equal chance of being in either of the treatment groups. The total study duration for the individual participants will be approximately one year.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine eligibility for the study
* Male or female, age more than or equal to 18 years at the time of signing informed consent
* Body mass index (BMI) more than or equal 30 kg/m^2
* Enrolled in Cleveland Clinic Employee Health Plan, and expecting to be covered by the Cleveland Clinic Employee Health Plan for the duration of the study

Exclusion Criteria:

* Contraindications to all of the medications approved by the FDA for chronic weight management according to the label
* Previous participation in this study. Participation is defined as signed informed consent
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)
* Participation in another clinical trial within 30 days before screening
* Treatment with any medication with the intention of weight loss within 90 days before screening
* Previous or current participation in Cleveland Clinic's Integrated Medical Weight Management Program
* History of (or plans during the study period for) bariatric surgery, or use of minimally-invasive weight loss devices (i.e. Intragastric balloons, lap bands) not removed within 1 year prior to screening
* History of type 1 or type 2 diabetes mellitus
* Hemoglobin A1c (HbA1c) more than or equal to 6.5% at screening or within 90 days prior to randomization
* Any condition, unwillingness or inability, not covered by any of the other exclusion criteria, which, in the study clinician's opinion, might jeopardize the subject's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com

REFERENCES:
- [Derived] Pantalone KM, Rogen B, Zirm P, Xiao H, Bena J, Barnard G, Borukh E, Peechakara S, Griebeler ML, Young JB, Burguera B. An Obesity-Centric Approach with and Without Anti-Obesity Medications Compared to the Usual-Care Approach to Management of Patients with Obesity and Type 2 Diabetes in an Employer Setting: A Pragmatic Randomized Controlled Trial (EMPOWER-T2D). Diabetes Ther. 2024 May;15(5):1201-1214. doi: 10.1007/s13300-024-01563-0. Epub 2024 Apr 4. PMID 38573466
- [Derived] Pantalone KM, Smolarz BG, Ramasamy A, Baz Hecht M, Harty BJ, Rogen B, Griebeler ML, Borukh E, Young JB, Burguera B. Effectiveness of Combining Antiobesity Medication With an Employer-Based Weight Management Program for Treatment of Obesity: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2116595. doi: 10.1001/jamanetworkopen.2021.16595. PMID 34255049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at a single site in the United States.
Pre-assignment Details: Participants were randomized in a 1:1 manner to receive either Cleveland Clinic's Integrated Medical Weight Management Program (WMP) with medication for chronic weight management (WMP + Rx) or Cleveland Clinic's Integrated Medical WMP alone (WMP).
Groups:
- Weight Management Program (WMP) + Rx: Participants were to receive Cleveland Clinic's existing Integrated Medical WMP combined with medication for chronic weight management. Participants were prescribed any one of the 5 approved medicines: Xenical®, Belviq®, Qsymia®, Contrave® and Saxenda®.
- Weight Management Program (WMP): Participants were to receive Cleveland Clinic's existing Integrated Medical WMP.
Period: Overall Study
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Started | 100 | 100
Full Analysis Set (FAS) | 100 | 100
Completed | 96 | 91
Not Completed | 4 | 9
Not completed — Lost to Follow-up | 4 | 8
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP) | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.43) | 49.1 (10.11) | 50.0 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 89 | 177
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 96 | 100 | 196
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 80 | 66 | 146
    Black or African American | 19 | 33 | 52
    Asian/White | 1 | 0 | 1
    India | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Percentage change in body weight from baseline (month 0) to month 12 is presented.
Time Frame: Month 0, month 12
Population: The FAS comprised of all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Percent change of body weight
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 100 | 100
Percent change of body weight | -7.69 (0.72) | -4.19 (0.73)
Statistical Analysis 1: Comparison: Weight Management Program (WMP) + Rx vs Weight Management Program (WMP); Analysis of in-trial data with missing observations for body weight at month 12 imputed from the WMP arm based on a jump to reference multiple (x=100) imputation approach. Percent change in body weight from baseline to month 12 was calculated for each study participant within the FAS and analyzed using an analysis of covariance model with randomized treatment as a factor and baseline body weight (kg) as a covariate; Test type: Superiority; p < 0.001, ANCOVA; Treatment Difference = -3.50, 95% CI 2-sided [-5.51 to -1.50], Standard Error of Mean 1.02

2. Secondary Outcome: Participants Achieving 5% or More Reduction in Body Weight
Description: The percentage of participants achieving 5% or more reduction in body weight was analyzed using a logistic regression model with treatment as categorical effect and baseline weight (kg) as covariate. Percentage of participants who achieved 5% or more reduction in body weight from baseline at month 12 is presented.
Time Frame: Month 12
Population: The FAS comprised of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 100 | 100
Percentage of participants | 62.5 | 44.8

3. Secondary Outcome: Participants Achieving 10% or More Reduction in Body Weight
Description: The percentage of participants achieving 10% or more reduction in body weight was analyzed using a logistic regression model with treatment as categorical effect and baseline weight (kg) as covariate. Percentage of participants who achieved 10% or more reduction in body weight from baseline at month 12 is presented.
Time Frame: Month 12
Population: The FAS comprised of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 100 | 100
Percentage of participants | 34.7 | 22.4

4. Secondary Outcome: Number of Shared Medical Appointments (SMAs) Attended
Description: Shared medical appointments (SMAs) is a concept that combines group appointments for participants with clinical intervention, consisting of encounters with a nutritionist, exercise physiologist, and endocrinologist/obesity medicine specialist. The mean number of SMAs attended by the participants are presented.
Time Frame: Months 0-12
Population: The FAS comprised of all randomized participants.
Measure: Mean (Standard Deviation); unit: SMAs
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 100 | 100
SMAs | 9.7 (2.98) | 7.4 (3.90)

5. Secondary Outcome: Participants Attending 9 or More SMAs
Description: Shared medical appointment (SMA) is a concept that combines group appointments for participants with clinical intervention, consisting of encounters with a nutritionist, exercise physiologist, and endocrinologist/obesity medicine specialist. Number of participants who attended 9 or more SMAs is presented.
Time Frame: Months 0-12
Population: The FAS comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 100 | 100
Participants | 79 | 51

6. Secondary Outcome: Proportion of Days Covered by Prescription Claims for Medication for Chronic Weight Management
Description: Participants who enrolled in the WMP + Rx arm were provided a prescription for medication indicated for chronic weight management. Proportion of days covered by prescription claims for medication for chronic weight management is presented. This endpoint is applicable only for treatment arm, WMP + Rx.
Time Frame: Months 0-12
Population: The FAS comprised of all randomized participants.
Measure: Mean (Standard Deviation); unit: Proportion of days
Arm/Group | Weight Management Program (WMP) + Rx
Number analyzed (Participants) | 100
Proportion of days | 66.48 (27.096)

7. Secondary Outcome: Participants Covered by Prescription Claims for Medication for Chronic Weight Management for at Least 80% of Days
Description: Participants who enrolled in the WMP + Rx arm were provided a prescription for medication indicated for chronic weight management. Number of participants covered by prescription claims for medication for chronic weight management for at least 80% of days is presented. This endpoint is applicable only for treatment arm, WMP + Rx.
Time Frame: Months 0-12
Population: The FAS comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Management Program (WMP) + Rx
Number analyzed (Participants) | 100
Participants | 43

8. Secondary Outcome: Change in 'At-Work Productivity Loss Index' as Measured by Work Limitations Questionnaire Self-administered Short-Form (WLQ-8)
Description: The WLQ-8 questionnaire assesses the degree to which participants have difficulty related to time management, physical tasks, mental/interpersonal tasks, and output tasks due to their physical and/or emotional health. The WLQ-8 produces subscale scores as well as an index of overall at-work productivity loss. WLQ-8 outcomes are expressed as proportion time with difficulty, with higher scores indicating greater limitations, i.e., worse outcomes. The score ranges from 1 to 5 where '1' represents none of the time and, '5' represents all of the time. Change in 'At-Work Productivity Loss Index' from month 0 to month 12 is presented.
Time Frame: Month 0, month 12
Population: The FAS comprised of all randomized participants. Overall number of participants analyzed=number of participants contributed to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 100 | 98
Score on a scale | -0.06 (0.06) | -0.03 (0.06)

9. Secondary Outcome: Change in 'Time Management' as Measured by WLQ-8
Description: The WLQ-8 questionnaire assesses the degree to which participants have difficulty related to time management, physical tasks, mental/interpersonal tasks, and output tasks due to their physical and/or emotional health. WLQ-8 outcomes are expressed as proportion time with difficulty, with higher scores indicating greater limitations, i.e., worse outcomes. The score ranges from 1 to 5 where '1' represents none of the time and, '5' represents all of the time. Change in 'time management' from month 0 to month 12 is presented.
Time Frame: Month 0, month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 98 | 95
Score on a scale | -0.10 (0.07) | -0.19 (0.07)

10. Secondary Outcome: Change in 'Physical Tasks' as Measured by WLQ-8
Description: The WLQ-8 questionnaire assesses the degree to which participants have difficulty related to time management, physical tasks, mental/interpersonal tasks, and output tasks due to their physical and/or emotional health. WLQ-8 outcomes are expressed as proportion time with difficulty, with higher scores indicating greater limitations, i.e., worse outcomes. The score ranges from 1 to 5 where '1' represents none of the time and, '5' represents all of the time. Change in 'physical tasks' from month 0 to month 12 is presented.
Time Frame: Month 0, month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 99 | 98
Score on a scale | -0.09 (0.11) | -0.05 (0.11)

11. Secondary Outcome: Change in 'Mental/Interpersonal Tasks' as Measured by WLQ-8
Description: The WLQ-8 questionnaire assesses the degree to which participants have difficulty related to time management, physical tasks, mental/interpersonal tasks, and output tasks due to their physical and/or emotional health. WLQ-8 outcomes are expressed as proportion time with difficulty, with higher scores indicating greater limitations, i.e., worse outcomes. The score ranges from 1 to 5 where '1' represents none of the time and, '5' represents all of the time. Change in 'mental/interpersonal tasks' from month 0 to month 12 is presented.
Time Frame: Month 0, month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 98 | 97
Score on a scale | -0.06 (0.09) | -0.03 (0.09)

12. Secondary Outcome: Change in 'Output Tasks' as Measured by WLQ-8
Description: The WLQ-8 questionnaire assesses the degree to which participants have difficulty related to time management, physical tasks, mental/interpersonal tasks, and output tasks due to their physical and/or emotional health. WLQ-8 outcomes are expressed as proportion time with difficulty, with higher scores indicating greater limitations, i.e., worse outcomes. The score ranges from 1 to 5 where '1' represents none of the time and, '5' represents all of the time. Change in 'output tasks' from month 0 to month 12 is presented.
Time Frame: Month 0, month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 97 | 98
Score on a scale | 0.07 (0.10) | 0.12 (0.11)

13. Secondary Outcome: Change in 'Absenteeism: Percent Work Time Missed Due to Excess Weight' as Measured by Work Productivity and Activity Impairment Questionnaire Specific Health Problem V2.0 (WPAI:SHP)
Description: The WPAI:SHP questionnaire assesses both work productivity through absenteeism (i.e., work time missed), presenteeism (i.e., impairment at work or reduced on-the-job effectiveness), and work productivity loss, as well as daily activity impairment (e.g., work around the house, shopping, exercising, childcare, studying) attributable to excess weight. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity. Negative numbers indicate improvement from baseline.
Time Frame: Month 0, month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 95 | 95
Score on a scale | -0.43 (0.17) | -0.48 (0.19)

14. Secondary Outcome: Change in 'Presenteeism: Percent Impairment While Working Due to Excess Weight' as Measured by WPAI:SHP
Description: as for outcome 13
Time Frame: Month 0, month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 95 | 95
Score on a scale | -1.88 (1.62) | -1.94 (1.82)

15. Secondary Outcome: Change in 'Work Productivity Loss: Percent Overall Work Impairment Due to Excess Weight' as Measured by WPAI:SHP
Description: as for outcome 13
Time Frame: Month 0, month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 95 | 95
Score on a scale | -1.84 (1.62) | -1.89 (1.82)

16. Secondary Outcome: Change in 'Percent Activity Impairment Due to Excess Weight' as Measured by WPAI:SHP
Description: as for outcome 13
Time Frame: Month 0, month 12
Population: The FAS comprised of all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
Number analyzed (Participants) | 100 | 100
Score on a scale | -9.95 (2.53) | -7.20 (2.69)

ADVERSE EVENTS:
Time Frame: Months 0 - 12
Description: All study medications used in this study were approved for the treatment of chronic weight management at the time of their use and prescribed at the discretion of the study clinician according to routine practice. For this reason, only SAEs and pregnancies (in female participants) were collected.
Arm/Group | Weight Management Program (WMP) + Rx | Weight Management Program (WMP)
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/100
Serious Adverse Events (participants affected / at risk) | 8/100 | 11/100
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Management Program (WMP) + Rx (N=100) | Weight Management Program (WMP) (N=100)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis Salmonella (Gastrointestinal disorders) | 0 (0) | 1 (1)
Procedural Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plasma Cell Myeloma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Ovarian Mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Organ Donor (Social circumstances) | 1 (1) | 0 (0)
Gastric Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Dizziness (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03799198/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03799198/SAP_001.pdf